CLINICAL TRIAL: NCT04776239
Title: Allogeneic Mesenchymal Human Stem Cell Infusion Therapy for Endothelial DySfunctiOn in Diabetic Subjects With Symptomatic Ischemic Heart Disease.
Brief Title: Allogeneic Mesenchymal Human Stem Cell Infusion Therapy for Endothelial DySfunctiOn in Diabetic Subjects With Symptomatic Ischemic Heart Disease. (ACESO-IHD)
Acronym: ACESO-IHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua M Hare (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Professor of Clinical Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200874; 1R01HL134558-01 (NIH)
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus; Ischemic Heart Disease
Keywords: Endothelial dysfunction; Diabetes; Stem cells
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Allogeneic Mesenchymal Stem Cells (MSCs) Group (Experimental): Participants in this group will be receive a single administration of intravenous allogeneic human Mesenchymal Stem Cells (hMSCs) (100 million).
  Interventions: Drug: 100 million Allogeneic Mesenchymal Human Stem Cells
- Group 2: Placebo Group (Experimental): Participants in this group will receive a single dose of placebo (Cell-free PlasmaLyte-A medium supplemented with 1% HSA) infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 100 million Allogeneic Mesenchymal Human Stem Cells — 1 single intravenous infusion
  Other Names: allo-human Mesenchymal Stem Cells (hMSCs); stem cells
  Arms: Group A: Allogeneic Mesenchymal Stem Cells (MSCs) Group
Other: Placebo — Placebo delivered via peripheral intravenous infusion
  Arms: Group 2: Placebo Group

SUMMARY:
The purpose of this study is to test the hypothesis that allogeneic Mesenchymal Stem Cells (MSCs) promote systemic and coronary endothelial repair through rescue of bone marrow progenitors in type 2 diabetic patients with symptomatic IHD compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age (males and females).
2. Provide written informed consent.
3. Have a diagnosis of symptomatic ischemic heart disease (IHD) and an indication for standard-of-care coronary angiography.
4. Have Diabetes Mellitus (DM) type 2 documented by glycated hemoglobin (HbA1C) > 7%, or on medical therapy for diabetes.

Exclusion Criteria:

1. Be younger than 18 years of age.
2. Have history of prior myocardial Infarction and revascularization.
3. Have a baseline glomerular filtration rate (GFR) <30 ml/min 1.73m2 estimated using the Modification of Diet for Renal Disease (MDRD) formula.
4. Have poorly controlled blood glucose levels with hemoglobin A1C > 8.5% in the previous 3 months.
5. Have a history of proliferative retinopathy or severe neuropathy requiring medical treatment.
6. Have an indication for standard-of-care surgical (including valve surgery, placement of left-ventricular assist device) or percutaneous intervention for the treatment of valvular heart disease (including valvuloplasty).
7. Have known hypersensitivity or contraindication to aspirin; both heparin and bivalirudin; all available P2Y12 inhibitors (clopidogrel, prasugrel, and ticagrelor); or any zotarolimus, cobalt, chromium, nickel, tungsten, acrylic, or fluoropolymers; or hypersensitivity to contrast media that cannot be adequately premedicated.
8. Have a hematologic abnormality as evidenced by hematocrit < 25%, white blood cell < 2,500/microliter (uL) or platelet values < 100,000/uL without another explanation (per investigator discretion).
9. Have liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the upper limit of normal.
10. Have a bleeding diathesis or coagulopathy (INR > 1.3), cannot be withdrawn from anticoagulation therapy, or will refuse blood transfusions.
11. Be an organ transplant recipient or have a history of organ or cell transplant rejection.
12. Have a clinical history of malignancy within the past 5 years (i.e., subjects with prior malignancy must be disease free for 5 years), except curatively-treated basal cell or squamous cell carcinoma, or cervical carcinoma.
13. Have a condition that limits lifespan to < 1 year.
14. Have a history of drug or alcohol abuse within the past 24 months.
15. Be serum positive for HIV, hepatitis B surface antigen (sAg), or viremic hepatitis C.
16. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
17. Be pregnant, nursing, or of childbearing potential and not on contraceptive medications. (May participate if on 2 forms of contraceptives).
18. Any other condition that in the judgment of the Investigator would be a contraindication to enrollment or follow-up.
19. Coronary lesions with restenosis or heavy calcification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
EPC-CFU levels | 6 months post-infusion
  Endothelial progenitor cells (EPC)-colony forming units (CFUs) will be assessed from blood samples. The unit of measure is the average number of colonies per well.
Flow Mediated Diameter Percentage (FMD%) | 6 months post-infusion
  FMD% is measured via brachial artery ultrasound. The unit of measure is percent.

SECONDARY OUTCOMES:
Target lesion lumen loss | 6 months (post-infusion)
  Target lesion lumen loss as assessed by quantitative coronary angiography (QCA). The unit of measure is millimeters (mm).
Circulating angiogenic factors marker levels | 6 months post-infusion
  Circulating angiogenic marker levels will be assessed from blood samples. The unit of measure is pg/mL
Circulating inflammatory markers | 6 months post-infusion
  Circulating inflammatory markers including will be assessed from blood samples. The unit of measure is pg/mL.
Seattle Angina Questionnaire (SAQ) Angina Frequency | 6 months post-infusion
  SAQ is a 7 item questionnaire with a total score ranging from 0-100 with the higher scores indicating less physical limitations, less angina, symptom frequency and better quality of life. The unit of measure is score on a scale.
EuroQol 5 Dimension (EQ-5D) Quality of life Questionnaire Overall Health Status Question | 6 months post-infusion
  EQ-5D Quality of Life Questionnaire Overall Health Status question has a total score ranging from 0-100 with higher scores indicating better quality of life. The unit of measure is score on a scale.
Short Form (SF) 36 Questionnaire Quality of Life Questionnaire | 6 months post-infusion
  SF 36 Quality of Life Questionnaire consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a score on an scale of 0-100. Lower scores indicate the more disability, and higher scores indicate less disability.
Number of Treatment-Emergent Serious Adverse Events (TE-SAE) | 1 month post infusion
  TE-SAEs will be defined as the composite of: death, non-fatal myocardial infarction (MI), stroke, hospitalization for heart failure, sustained ventricular arrhythmias (characterized by ventricular arrhythmias lasting longer than 30 sec or with hemodynamic compromise) or atrial fibrillation at 1 month post-infusion. TE-SAEs will be assessed by treating physician. The unit of measure is number of events.
Number of Major Adverse Cardiac Events (MACE) | 12 months
  Defined as the composite incidence of (1) death, (2) hospitalization for cardiovascular events or (3) non-fatal myocardial infarction MI at 1 year. MACE will be assessed by treating physician. The unit of measure is number of events
Number of Treatment Emergent Adverse Events | 12 months
  Rates of treatment emergent adverse event (AE) as assessed by treating physician will be reported. The unit of measure is number of events.
Number of participants with abnormal lab values | 12 months
  Number of participants with clinically significant abnormal serum hematology and clinical chemistry values will be reported. Clinical significance will be assessed by treating physician. The unit of measure is number of participants.
Number of participants with Target Vessel Failure | 12 months
  Number of participants with target vessel failure will be reported. Target vessel failure is defined as any participant that encounters revascularization, death, or MI attributed to the target vessel post-PCI. The unit of measure is number of participants.
Post-Percutaneous Coronary Intervention (PCI) coronary artery endothelial function as assessed via CFR | 6 months (post-infusion)
  Coronary Flow Reserve (CFR) as measured via cardiac catheterization angiography. The value is expressed as a ratio that is calculated by dividing the maximum coronary blood flow (mL/min/g) by the resting blood flow (mL/min/g)
Post-PCI coronary artery endothelial function as assessed via FFR | 6 months (post infusion)
  Fractional Flow Reserve (FFR) as measured via cardiac catheterization angiography. FFR is a dimensionless number that ranges from 0 to 1 that is a ratio of two pressures (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Spilias, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description: Interdisciplinary Stem Cell Institute at the University of Miami Miller School website — http://isci.med.miami.edu